CLINICAL TRIAL: NCT05897892
Title: School of Environmental Sciences - University of Indonesia
Brief Title: The Clinical Study on the Mangrove Sword Bean Food Bar Effect for Older People
Acronym: FF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Fatmah Fatmah, Principal Investigator, Indonesia University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SILUI
Record Dates: First submitted 2023-05-23; First posted 2023-06-09 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Nutrition Disorders in Old Age; Disaster
Keywords: Older people; disaster; weight; mangrove-sword bean food bar
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Intervention Model Description: Treatment group consumed mangrove sword bean food bar during 15 days. Control group consumed sword bean food bar during 15 days. Balanced nutrition education undertaken to all subjects at two groups once at the first week of study.
Who Masked: Participant
Masking Description: Treatment group consumed mangrove sword bean food bar during 15 days. Control group consumed sword bean food bar during 15 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Treatment group received 50 g mangrove sword bean food bar each day during 15 days.
  Interventions: Dietary Supplement: Clinical study on the mangrove sword bean food bar effect for older people
- Control Group (Placebo Comparator): Control group received 50 g sword bean food bar per day during 15 days.
  Interventions: Dietary Supplement: Clinical study on the mangrove sword bean food bar effect for older people

INTERVENTIONS:
Dietary Supplement: Clinical study on the mangrove sword bean food bar effect for older people — The treatment group consumed 50 g mangrove sword bean food bar each day during 15 days.
  Other Names: EFP

SUMMARY:
The goal of this clinical study is to assess the api-api mangrove sword bean food bar effect on the older people's weight affected by a landslide

The main questions aimed to answer are:

* Can api-api mangrove sword bean food bar improve the weight of older people affected by landslide?
* Can balanced nutrition education increase the older peoples' knowledge?

Participants divided in the two groups i.e.:

* Treatment group received 50 g mangrove sword bean food bar each day during 15 days.
* Control group received 50 g sword bean food bar each day during 15 days.
* Both groups obtained balanced nutrition of older people education once at the first week of study.

DETAILED DESCRIPTION:
Treatment group received 50 g mangrove sword bean food bar each day during 15 days.

Control group received 50 g sword bean food bar each day during 15 days. Both groups obtained balanced nutrition of older people education once at the first week of study.

Compliance monitoring to control the food compliance by the subjects at two groups through home visit, weight measurement, three days food recall, and food bar distribution checking by trained enumerators.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years old or above
* Male and female
* Living in Cihanjuang Village, Sumedang District, West Java Province Indonesia who affected by the landslide disaster
* Had normal, under-, or over-nutrition status
* Not suffering from chronic diseases or degenerative diseases during the study.
* Willing to avoid consumption of any snacks other than the food bars and plain water.

Exclusion Criteria:

* Having difficulty mobilities to run daily basic activities.
* Suffered from infectious and or a chronical diseases.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
Mangrove sword bean food bar on the weight of older people | Two weeks
  50 g mangrove sword bean food bar each day given to treatment group. 50 g sword bean food bar each day consumed by the control group. Weight measured by digital weighing SECA by trained enumerator at the first week and the second week of study.

SECONDARY OUTCOMES:
Balanced nutrition knowledge of older people | Two weeks
  Both groups received the balance nutrition education once at the second week of study.
  The knowledge change of older people measured by the baseline and end-line questionnaires by trained enumerators

CONTACTS AND LOCATIONS:
Overall Officials: Fatmah Fatmah, Dr., Principal Investigator — Indonesia University
Locations (1):
- Health integrated post for older people office, Sumedang, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fatmah F. Effectiveness of mangrove sword bean food bar addressed to older people of landslide disaster victims. Front Nutr. 2024 Apr 8;11:1291580. doi: 10.3389/fnut.2024.1291580. eCollection 2024. PMID 38650640